CLINICAL TRIAL: NCT03343782
Title: Outcomes of Expanded Autologous Bone Marrow-derived Mesenchymal Stem Cells Therapy in Type 2 Diabetes
Brief Title: Outcomes of Expanded Autologous Bone Marrow-derived Mesenchymal Stem Cells Therapy in Type II Diabetes
Acronym: ASD2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VinmecRISCGT70
Record Dates: First submitted 2017-11-12; First posted 2017-11-17 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes; BM mesenchymal stem cell
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cell transplantation (Experimental): Intervention: 30 patients will be transplanted autologous bone marrow-derived mesenchymal stem cells and undergoing 2 treatment with 6 months interval
  Interventions: Combination Product: Expanded autologous bone marrow-derived mesenchymal stem cell

INTERVENTIONS:
Combination Product: Expanded autologous bone marrow-derived mesenchymal stem cell — Collect bone marrow from lilac crest using local anaesthetic and syringe collection. Mesenchymal stem cell will be isolated, expanded and characterized in vitro under the GMP- grade procedure

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of autologous bone marrow-derived mesenchymal stem cells transplantation in the treatment of type 2 diabetes mellitus

DETAILED DESCRIPTION:
Bone marrow-derived mesenchymal stem cells have the immunosuppressive effect and secrete a variety of cytokines, improve the microenvironment of diabetic patients, targeting insulin resistance tissue, ameliorate the metabolic disorder of islet damage, protect and regeneration of the islet beta cells; reduce high blood sugar.The purpose of this study is to evaluate the safety and effectiveness of autologous bone marrow-derived mesenchymal stem cells transplantation in treatment 30 patients with type 2 diabetes mellitus at Vinmec International Hospital, Hanoi, Vietnam

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age from 18 years and above.
* Hemoglobin A1c (HbA1c) is ranged from 7.5% to 9% at baseline.
* Type 2 diabetes duration 5 years or more.
* Before the screening, joint or combined with insulin, oral medications to treat more than 3 months.
* Who signed the informed consent form.

Exclusion Criteria:

* Type 1 diabetes.
* Chronic disease or severe disease, including cancer, severe heart disease, kidney disease, liver disease, etc.
* According to the medical doctor's judgement, may endanger the safety of the subjects

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Insulin dose | up to the 12-month period following treatment
  Reduction of insulin dose requirement by ≥50% in both groups
Adverse events | up to the 12-month period following treatment
  Number of adverse events in both groups

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) level | up to the 12-month period following treatment
  Improvement of HbA1c level as compared to baseline between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nguyen LT, Hoang DM, Nguyen KT, Bui DM, Nguyen HT, Le HTA, Hoang VT, Bui HTH, Dam PTM, Hoang XTA, Ngo ATL, Le HM, Phung NY, Vu DM, Duong TT, Nguyen TD, Ha LT, Bui HTP, Nguyen HK, Heke M, Bui AV. Type 2 diabetes mellitus duration and obesity alter the efficacy of autologously transplanted bone marrow-derived mesenchymal stem/stromal cells. Stem Cells Transl Med. 2021 Sep;10(9):1266-1278. doi: 10.1002/sctm.20-0506. Epub 2021 Jun 3. PMID 34080789